CLINICAL TRIAL: NCT06911580
Title: Investigation of the Immediate Effects of Graston Massage on Muscle Mechanical Properties and Sports Performance in Elite Female Handball Players With Isolated Gastrocnemius Tightness
Brief Title: Immediate Effects of Graston Massage on Muscle Properties and Performance in Elite Female Handball Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Giresun University (Other)
Responsible Party: Principal Investigator, Nihat Sarıalioğlu, Assistant Professor, Giresun University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GRU-SBF-NS-03
Record Dates: First submitted 2025-03-24; First posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Isolated Gastrocnemius Tightness
Keywords: handball; graston; Isolated gastrocnemius tightness; Muscle mechanical properties; Performance

STUDY DESIGN:
Intervention Model Description: The study was designed as a quasi-experimental research.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Physical Tests and Measurements (Other): Assessment of Muscle Mechanical Properties:The Myoton PRO muscle palpation device was used for the evaluation.
  Strength Measurement: Strength measurement was performed on the calf muscle group. The Activforce Digital Dynamometer, which has been reported to have a high level of reliability, was used for this assessment.
  Agility Test:Agility values were determined using the Illinois Agility Test, measured with a photocell electronic stopwatch system with a precision of 0.01 seconds. The test was conducted twice, and the best result was recorded.
  Vertical Jump Test:Vertical jump values were measured using a Smart Speed electronic jump mat with the hands-free (arm swing) countermovement jump technique. The athlete positioned themselves with their feet shoulder-width apart on the jump mat.
  Interventions: Procedure: Graston Massage

INTERVENTIONS:
Procedure: Graston Massage — The participant was positioned prone on the treatment table with the knee slightly flexed. A small amount of lubricating gel was applied to the entire gastrosoleus complex and the calcaneal tendon. For one minute, sweeping strokes were performed downwards on the gastrocnemius heads using the GT-5 tool. From the second to the fourth minute, the GT-5 was used in an upward direction to ensure that both the gastrocnemius and soleus were treated. Afterward, with the GT-2 tool, one minute of downward sweeping and one minute of upward sweeping were performed on the calcaneal tendon. Following the two minutes of sweeping, GT-3 was used to apply short, perpendicular strokes to the medial and lateral sides of the calcaneal tendon, with 30 seconds for each side. The total application lasted approximately 7 minutes (Palmer et al., 2017).

SUMMARY:
The aim of this study is to investigate the immediate effects of Graston massage on muscle mechanical properties and sports performance in elite handball players with isolated gastrocnemius tightness.

DETAILED DESCRIPTION:
Handball is a high-paced competitive sport that requires advanced physical demands. The ability to achieve the desired performance in handball is influenced by the functionality of the lower extremities. One of the key structures responsible for the mobility of the lower extremities is the gastrocnemius muscle. The gastrocnemius is a superficial, two-headed skeletal muscle located in the posterior part of the leg, with its primary function being plantar flexion of the ankle. Due to intense usage, improper training models, or various traumas, structural abnormalities may develop in the gastrocnemius muscle among athletes. One of the most common structural disorders is isolated gastrocnemius tightness (IGT). IGT is considered critical in terms of sports injuries and performance and is also recognized as a prevalent disorder even in the general population.

IGT, which arises as a result of gastrocnemius-soleus contracture, is a muscle dysfunction characterized by increased stiffness of the ankle joint in dorsiflexion. Restrictions in dorsiflexion caused by IGT can increase pressure on soft tissues during changing conditions and sudden movements in training and competitions, leading to a higher risk of injury and potential declines in sports performance. Chronic muscle tightness also affects the viscoelastic properties of the muscle. Mechanical muscle properties such as muscle tone and stiffness are considered fundamental elements for maintaining efficient muscle contractions in terms of both function and energy. A shortened and tight skeletal muscle may hinder potential force production, leading to increased muscle tone and stiffness. Increased tone and stiffness, in turn, can reduce movement efficiency and contribute to a higher risk of injuries.

IGT can be alleviated through various interventions, including exercise models, surgical procedures, and myofascial release techniques. The Graston technique is recommended for restoring optimal length in the myofascial complex, enhancing function, and improving hypomobility caused by skeletal muscle tightness.

Previous studies have emphasized the importance of IGT and its treatment. However, no comprehensive study has been found regarding the effects of preventive measures against IGT on sports performance and muscle properties in athletes. Identifying IGT and implementing effective compensatory mechanisms play a crucial role in maintaining athlete health and sustaining performance, highlighting the significance of this research.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have IGT in at least one leg.
* Age range must be between 19-27 years.
* Must have been a licensed handball player for at least the past five years.
* Must not have undergone any surgical operation in the past year.

Exclusion Criteria:

* Participants who are in their menstrual period will be excluded from the study.
* Those who have used pharmacological products classified as muscle relaxants or derivatives within the last 24 hours will be excluded.
* Those who do not meet the inclusion criteria will be excluded from the study.

Ages: 19 Years to 27 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-02-20 (Actual)

PRIMARY OUTCOMES:
IGT (isolated gastrocnemius tightness) Assessment | Baseline
  The Silfverskiold test was used to identify gastrocnemius tightness, which is characterized by an equinus deformity at the ankle when the knee is extended but disappears when the knee is flexed. In this test, gastrocnemius equinus is determined when passive ankle dorsiflexion is ≤5 degrees with the knee fully extended, but increases to ≥15 degrees when the knee is flexed to 90 degrees. Participants were positioned supine on a treatment table, and goniometric measurements were taken according to the test protocol. Those who met the Silfverskiold criteria in at least one leg were classified as having IGT. (physiological parameter)
Assessment of Muscle Mechanical Properties | Baseline
  The Myoton PRO muscle palpation device was used for the evaluation. Myoton PRO is a portable, non-invasive device with established reliability and objectivity in assessing muscle mechanical properties. The device consists of a body and a probe. The probe applies mechanical pressure to the surface, generating a rapid deformation through a mechanical impulse. This deformation induces damped natural oscillations in the soft tissue, which are recorded by an accelerometer. During the application, the participant was positioned supine on a treatment table. To ensure the most relaxed position of the muscle, a small cushion was placed under the tibia, supporting the ankle. Following the device protocol, three impulses were applied to the reference point of the medial gastrocnemius using the probe. All measurements were performed by the same expert physiotherapist. (physiological parameter)
Measuring Strength | Baseline
  Strength measurement was performed on the calf muscle group. The Activforce Digital Dynamometer, which has been reported to have a high level of reliability, was used for this assessment. The device was fixed to the wall at foot level, and the participant, lying in a supine position, was instructed to apply maximum plantar flexion force against it. To prevent any backward movement that could affect the measurement, support was provided to the participant at the shoulder region during the test. (physiological parameter)
Measuring Agility | Baseline
  Agility values were determined using the Illinois Agility Test, measured with a photocell electronic stopwatch system with a precision of 0.01 seconds. The test was conducted twice, and the best result was recorded. (physiological parameter)
Vertical Jump Test | Baseline
  Vertical jump values were measured using a Smart Speed electronic jump mat with the hands-free (arm swing) countermovement jump technique. The athlete positioned themselves with their feet shoulder-width apart on the jump mat. Once ready, the athlete bent down and jumped vertically to the highest point they could reach, landing back on the mat. Three trials were performed in the correct position, with a 3-second rest between each jump, and the best result was recorded in centimeters. Jumps were repeated with the knees flexed while the athlete was airborne. (physiological parameter)

CONTACTS AND LOCATIONS:
Locations (1):
- Giresun University, Giresun, Centre, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I don't want my data to be shared.